CLINICAL TRIAL: NCT01275027
Title: A Phase II, Placebo-Controlled, Randomized, Safety and Efficacy Study to Evaluate the Change in Hemoglobin A1c Levels in Type 2 Diabetic Subjects While Taking Nutralin
Brief Title: A Placebo-Controlled, Randomized, Safety and Efficacy Study to Evaluate the Change in Hemoglobin A1c Levels in Type 2 Diabetic Subjects While Taking Nutralin
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor recalled the study
Sponsor: Avera McKennan Hospital & University Health Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ARI-1340-Nutralin
Record Dates: First submitted 2011-01-10; First posted 2011-01-12 (Estimated); Last update posted 2015-04-22 (Estimated); Status verified 2015-04

CONDITIONS: Diabetes
Keywords: diabetes; blood sugar; insulin; nutritional supplement; nutraceutical
MeSH Terms: conditions — Diabetes Mellitus; Insulin Resistance

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Nutralin (Experimental): Individuals with Type 2 Diabetes
  Interventions: Dietary Supplement: Nutralin
- Placebo (Placebo Comparator): Individuals with Type 2 Diabetes
  Interventions: Dietary Supplement: Nutralin

INTERVENTIONS:
Dietary Supplement: Nutralin — 7 capsules taken 15 minutes before each of the three main meals of the day

SUMMARY:
The purpose of this clinical research study is to evaluate the effects an investigational food product has on the blood sugar and insulin levels in individuals with diabetes.

DETAILED DESCRIPTION:
The investigational product has helped decrease the amount of insulin needed in treating diabetic dogs and has improved the dogs' longevity and quality of life. Observational analysis by trained veterinarians has indicated that the natural fluctuations in blood glucose levels do not exist in dogs consuming the product. An initial Phase 1 study tested the product in a brownie form. The product has been reformulated to capsule form for the Phase 2 study.

The hypothesis for this study is that diabetic individuals will decrease their insulin/diabetic medication usage and have a decrease in glucose levels after consuming the product for 16 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Men and women who are at least 18 years old
* Diagnosis of Type 2 Diabetes
* Has been on stable diabetes medication/insulin for the past three months

Exclusion Criteria:

* Women who are pregnant, breastfeeding or planning to become pregnant
* Diagnosis of Celiac Disease or gluten intolerance
* Current or active kidney disease
* Current or active liver disease
* Any food allergies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-01; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Blood Sugar | 16 weeks
  blood sugar levels
HgA1c reduction | 16 weeks
  reduction of Hemoglobin A1c levels

SECONDARY OUTCOMES:
Diabetes medication | 16 weeks
  reduction in the amount of diabetes medication needed

CONTACTS AND LOCATIONS:
Overall Officials: Edward Zawada, MD, Principal Investigator — Avera McKennan Hospital & University Health Center
Locations (1):
- Avera Research Institute, Sioux Falls, South Dakota, United States